CLINICAL TRIAL: NCT04836962
Title: Does the Single Use of Intravenous Dexamethasone Enhance Analgesic Quality of Pudendal Analgesia in Children Undergoing Hypospadias Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2021-0149
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Patients Undergoing Hypospadias Surgery
MeSH Terms: interventions — Saline Solution; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): normal saline is administrated to patients.
  Interventions: Drug: normal saline
- dexamethasone (Experimental): 0.5mg/kg dexamethasone is administered to patients.
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: normal saline — 2cc of normal saline is administered to patient instead of dexamethasone.
  Arms: control
Drug: dexamethasone — dexamethasone is administered 0.5mg/kg (up to 10mg) which is diluted with normal saline to make a total of 2cc.
  Arms: dexamethasone

SUMMARY:
Hypospadias is a congenital malformation that occurs in an embryological process, and occurs with an incidence of about 1/300 in male children. The caudal block was the most commonly performed method for pain control after hypospadias surgery, and showed very good analgesic effect in the immediate postoperative stage. However, the caudal block is a neuraxial block that has a limitation in its duration with single shot and shows complications and adverse effects. In recent studies, the pudendal nerve block has been suggested as an alternative method. In children undergoing hypospadias surgery, the pudendal nerve block showed a longer duration compared to the caudal block, decreased the use of analgesics within 24 hours after surgery, and showed higher parental satisfaction. On the other hand, there have been many studies to prolong the duration of the relatively short duration of caudal block. Among them, dexamethasone administered intravenously is known to improve the duration of various regional blocks and reduce the administration of additional analgesics. The aim of this study is to verify whether a single administration of dexamethasone can enhance the effect of the pudendal nerve block in children 0.5-3 years of age undergoing hypospadias surgery.

ELIGIBILITY:
Inclusion Criteria:

1. pediatric patients aged 6 months to 3 years who are planning to undergo hypospadias surgery
2. American Society of Anesthesiologists (ASA) classification 1~2

Exclusion Criteria:

1. patients who are having uncorrected heart deformity
2. patients who are having vertebrae deformity in which the pudendal nerve block cannot be performed
3. patients with blood coagulopathy
4. patients with diagnosed diabetes
5. patients with diagnosed adrenal disease
6. patients with fever above 37.5 degrees before surgery
7. patients currently taking steroids
8. patients contraindicated for dexamethasone administration

Ages: 6 Months to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
the duration from surgery to first PCA(patient-controlled analgesia) administration | during 48 hours after surgery
  the very first time of PCA usage after surgery, which is automatically recorded in PCA.

SECONDARY OUTCOMES:
the amount of additional analgesia required for postoperative 48hrs. | during 48 hours after surgery
  the amount of PCA usage for 48 hrs after surgery, which is automatically recorded in PCA.
the number of additional analgesia required for postoperative 48hrs. | during 48 hours after surgery
  the number of PCA usage for 48 hrs after surgery, which is automatically recorded in PCA.
pain score for each time period | during 48 hours after surgery
  ask parents about their children's pain score at each time point
overall parents' satisfaction questionnaire | 48 hours after surgery
  at 48 hours after surgery, parents are asked about satisfaction of their children's pain control

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Rim Lee, Principal Investigator — Department of Anesthesiology and Pain Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No